CLINICAL TRIAL: NCT01141452
Title: Retrospective, Real-life Evaluation of the Effectiveness, Cost-effectiveness and Direct Healthcare Costs of Qvar Pressurised Metered-dose Inhaler (pMDI) Compared With Beclometasone Dipropionate pMDI and Fluticasone pMDI in the Management of Chronic Obstructive Pulmonary Disease (COPD) in a Representative UK Primary Care Patient Population
Brief Title: Real-life Effectiveness and Cost-effectiveness of Qvar Versus FP and BDP in the Management of COPD
Acronym: QvarCOPD
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Professor David Price, Research in Real Life Limited
Other Study IDs: BA5
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; inhaled corticosteroid; increase; initiate; exacerbations; treatment success
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- IPDA FP MDI: Patients who were on inhaled corticosteroid therapy as part of their baseline therapy (any ICS therapy) who, at an index prescription date, stepped-up ICS dose as fluticasone via metered dose inhaler
  Interventions: Drug: Fluticasone propionate metred dose inhaler
- IPDA HFA-BDP MDI: Patients who were on inhaled corticosteroid therapy as part of their baseline therapy (any ICS therapy) who, at an index prescription date, stepped-up ICS dose as extra-fine hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler
  Interventions: Drug: Extra-fine hydrofluoroalkane beclomethasone MDI
- IPDA CFC-BDP MDI: Patients who were on inhaled corticosteroid therapy as part of their baseline therapy (any ICS therapy) who, at an index prescription date, stepped-up ICS dose as chlorofluorocarbon beclomethasone dipropionate via metered dose inhaler
  Interventions: Drug: Chlorofluorocarbon beclomethasone metered dose inhaler
- IPDI CFC-BDP MDI: Patients who were not receiving inhaled corticosteroid therapy as part of their baseline therapy but who, at an index prescription date, initiated ICS as chlorofluorocarbon beclomethasone dipropionate via metered dose inhaler
  Interventions: Drug: Chlorofluorocarbon beclomethasone dipropionate
- IPDI HFA-BDP MDI: Patients who were not receiving inhaled corticosteroid therapy as part of their baseline therapy but who, at an index prescription date, initiated ICS as hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler
  Interventions: Drug: Hydrofluoroalkane beclomethasone metred dose inhaler
- IPDI FP MDI: Patients who were not receiving inhaled corticosteroid therapy as part of their baseline therapy but who, at an index prescription date, initiated ICS as fluticasone propionate via metered dose inhaler
  Interventions: Drug: Fluticasone propionate metred dose inhaler

INTERVENTIONS:
Drug: Extra-fine hydrofluoroalkane beclomethasone MDI — Step-up in baseline BDP-equivalent ICS dose
  Other Names: Qvar®
  Groups: IPDA HFA-BDP MDI
Drug: Chlorofluorocarbon beclomethasone metered dose inhaler — Step-up in baseline BDP-equivalent ICS dose
  Groups: IPDA CFC-BDP MDI
Drug: Fluticasone propionate metred dose inhaler — Step-up in baseline BDP-equivalent ICS dose
  Groups: IPDA FP MDI
Drug: Fluticasone propionate metred dose inhaler — Initiation of ICS therapy
  Groups: IPDI FP MDI
Drug: Hydrofluoroalkane beclomethasone metred dose inhaler — Initiation of ICS therapy
  Other Names: Qvar®
  Groups: IPDI HFA-BDP MDI
Drug: Chlorofluorocarbon beclomethasone dipropionate — Initiation of ICS therapy
  Groups: IPDI CFC-BDP MDI

SUMMARY:
The objective of this study is to compare the effectiveness, cost-effectiveness and direct healthcare costs of managing chronic obstructive pulmonary disease (COPD) in primary care patients with evidence of COPD who either initiate inhaled corticosteroid (ICS) therapy, or have an increase in their ICS dose, as hydrofluoroalkane (HFA) beclometasone dipropionate (BDP) (hereafter Qvar®), CFC-BDP (hereafter BDP) and fluticasone propionate (FP) via pressurised metered-dose inhalers.

DETAILED DESCRIPTION:
Current asthma guidelines in the UK are underpinned by evidence derived from randomised controlled trials (RCTs). Although RCT data are considered the gold standard, patients recruited to asthma RCTs are estimated to represent less than 10% of the UK's asthma population. The poor representation of the asthma population is due to a number of factors, such as tightly-controlled inclusion criteria for RCTs. There is, therefore, a need for more representative RCTs and real-life observational studies to inform existing guidelines and help optimise asthma outcomes.

Short randomised trials have shown that Qvar is at least as effective as FP pMDI and as BDP pMDI at half the prescribed dose in patients with asthma. There is also evidence to suggest that, in adults, HFA formulation as used by Qvar (featuring BDP in solution rather than suspension) may achieve 10-fold higher deposition compared with CFC-BDP.4 Furthermore, deposition in the peripheral regions is higher compared with CFC-BDP and the fine-particle formulation also offers greater tolerance of poor co-ordination of breathing and inhaler actuation, resulting in lower oro-pharyngeal deposition compared with CFC-BDP.

Evidence of the efficacy of ICS monotherapy in COPD remains mixed at this time. While Qvar and ICS monotherapy use in the treatment of COPD is currently off-label, it occurs in clinical practice in two common scenarios:

1. before a diagnosis of COPD is made
2. unlicensed use as monotherapy, or in combination with long-acting bronchodilators

The study hypothesis, therefore, is that Qvar treatment in COPD may be associated with improved disease management and control (as assessed by effectiveness, cost-effectiveness and direct healthcare costs of managing COPD) compared with other commonly used ICS therapies, namely BPD and FP, by virtue of its improved deposition throughout the lungs and the small airways.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥40 years at index prescription date
* COPD diagnosis:

  * diagnostic code, and
  * ≥2 prescriptions for COPD therapy in baseline year (at different points in time)

    * For the ICS increase cohort (i.e. IPDA) ≥1 of these prescriptions must be for ICS therapy.
    * Commence ICS therapy at any time (even if before COPD diagnosis is made)

Exclusion Criteria:

- A diagnostic read code for any other chronic respiratory disease (except asthma)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care COPD patients who at an index prescription date either initiated ICS therapy as extrafine HFA-BDP, CFC-BDP or FP via MDI or had an increase in baseline BDP-equivalent ICS dose the index data as extrafine HFA-BDP, CFC-BDP or FP via MDI
Sampling Method: Non-Probability Sample
Enrollment: 815377 (Actual)
Dates: Start 2001-01; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Total number of exacerbations; exacerbation rate ratio; time to first after IPD | Two-year outcome period
  Where exacerbations are defined as:
  * Unscheduled hospital admissions / A&E attendances:*
    * For COPD (definite code) and
    * Lower respiratory tract infections (LRTI) treated with antibiotics
  * Acute use of oral steroids
  * Antibiotics use with a lower respiratory read code within a ±5-day window
COPD treatment success | Two-year outcome period
  * No recorded hospital attendance for COPD or respiratory related events (i.e. with a lower respiratory read code), including:
    * Admission
    * A&E attendance
    * Out of hours attendance
  * No exacerbations of COPD ("definite" plus "possible" prescriptions as defined above)
  * No consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics.

SECONDARY OUTCOMES:
COPD treatment success factoring in change in therapy | Two-year outcome period
  Defined as absence of:
  * Exacerbations; and/or
  * Increase in dose of inhaled steroid; and/or
  * Change in delivery device, and/or
  * Change in ICS
  * Use of additional therapy not received in baseline year, split by:
    * LABA
    * Theophylline
    * LTRAs.
COPD treatment success factoring in change in therapy unrelated to cost savings | Two-year outcome period
  Defined as absence of:
  * Exacerbations; and/or
  * Increase in dose of inhaled steroid; and/or
  * Use of additional therapy not received in baseline year, split by:
    * LABA
    * Theophylline
    * LTRAs.
Change in ICS dosing | Two-year outcome period
  Proportion of patients who:
  * Remained on the same ICS (and/or combination therapy) throughout the outcome period
  * Remained on the same ICS dose throughout the outcome period, but had another therapy added
  * Received an ICS dose increase and / or therapy added to their ICS during the outcome period.
Rate of hospitalisations | Two-year outcomes
  Where hospitalisations are defined as
  * Admissions and A&E coded as:
    * lower respiratory-related, or
    * for COPD
  * Admissions and A&E coded as:
    * lower respiratory-related, or
    * for COPD
    * admission attendance occurring within a ±7 day window of an LRTI treated with antibiotics.
SABA usage | Two-year outcome
  Average SABA daily dose, categorised as: 0mcg, >0-100mcg, >100-200mcg, >200-400mcg, >400-800mcg, >800mcg.
Mortality | Two-years
  * Respiratory mortality
  * All-cause mortality
Incidence of pneumonia | Two-year outcome
  * Unconfirmed (i.e. all unique patients with codes for pneumonia) AND
  * Confirmed:
    * chest X-ray within a month of a pneumonia diagnosis, or
    * hospitalisation within a month of a pneumonia diagnosis
Incremental cost effectiveness ratio | Two-year outcome
  Difference in costs (HFA-BDP the comparator) over difference in effectiveness (using primary outcome of exacerbations)
Cost of total healthcare treatment | Two-year outcome
  Costs for each intervention:
  * including ICS costs
  * excluding ICS costs
Costs for COPD treatment | Two-year outcome
  Costs of COPD treatment:
  * including ICS costs
  * excluding ICS costs

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof. MD, Principal Investigator — Company Director; Alison Chisholm, MSc, Study Director — Research Project Director
Locations (1):
- General Practice Research Database, London, London, United Kingdom

REFERENCES:
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Travers J, Marsh S, Caldwell B, Williams M, Aldington S, Weatherall M, Shirtcliffe P, Beasley R. External validity of randomized controlled trials in COPD. Respir Med. 2007 Jun;101(6):1313-20. doi: 10.1016/j.rmed.2006.10.011. Epub 2006 Nov 17. PMID 17113277
- [Background] Appleton SL, Adams RJ, Wilson DH, Taylor AW, Ruffin RE; North West Adelaide Cohort Health Study Team. Spirometric criteria for asthma: adding further evidence to the debate. J Allergy Clin Immunol. 2005 Nov;116(5):976-82. doi: 10.1016/j.jaci.2005.08.034. PMID 16275363
- [Background] Leach CL, Davidson PJ, Boudreau RJ. Improved airway targeting with the CFC-free HFA-beclomethasone metered-dose inhaler compared with CFC-beclomethasone. Eur Respir J. 1998 Dec;12(6):1346-53. doi: 10.1183/09031936.98.12061346. PMID 9877489
- [Background] Barber JA, Thompson SG. Analysis and interpretation of cost data in randomised controlled trials: review of published studies. BMJ. 1998 Oct 31;317(7167):1195-200. doi: 10.1136/bmj.317.7167.1195. PMID 9794854
- See also: Optimum Patient Care is the Research in Real Life's sister company (a social enterprise organisation) — http://www.optimumpatientcare.org